CLINICAL TRIAL: NCT07306260
Title: Multicenter Prospective Non-randomized Controlled Study of Ella Photodynamic Therapy for Cervical HSIL/CIN2
Acronym: PDT for CIN2
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Collaborators: Women's Hospital School Of Medicine Zhejiang University (Other); First People's Hospital of Hangzhou (Other); First Affiliated Hospital of Ningbo University (Network); Shaoxing People's Hospital (Other); Linping First People's Hospital (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2025-1382
Record Dates: First submitted 2025-12-14; First posted 2025-12-29 (Actual); Last update posted 2025-12-29 (Actual); Status verified 2025-12

CONDITIONS: HSIL, High Grade Squamous Intraepithelial Lesion; CIN 2; HPV (Human Papillomavirus)-Associated; Photodynamic Therapy (PDT)
Keywords: photodynamic therapy; High Grade Squamous Intraepithelial Lesion; human papillomavirus; loop electrosurgical excision procedure; efficacy
MeSH Terms: conditions — Squamous Intraepithelial Lesions; Papillomavirus Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ALA-PDT Group (Experimental): ALA-PDT treatment for cervical lesions 6 to 9 times
  Interventions: Procedure: ALA-PDT
- LEEP Group (Active Comparator): LEEP surgery for cervical lesions
  Interventions: Procedure: LEEP surgery

INTERVENTIONS:
Procedure: ALA-PDT — Apply 20% ALA gel for 3 hours, followed by red light irradiation, repeated every 7-14 days for a total of 6-9 sessions.
  Arms: ALA-PDT Group
Procedure: LEEP surgery — After anesthesia, cervical iodine staining was performed, followed by LEEP.
  Arms: LEEP Group

SUMMARY:
This study evaluates the efficacy and safety of ALA-PDT versus LEEP in treating cervical HSIL/CIN2, aiming to demonstrate non-inferiority in clinical efficacy.

DETAILED DESCRIPTION:
This study aims to conduct a multicenter, prospective, concurrent non-controlled clinical trial to evaluate the clinical efficacy of 5-aminolevulinic acid photodynamic therapy (ALA-PDT) compared with loop electrosurgical excision procedure (LEEP) in patients with high-grade squamous intraepithelial lesion (HSIL/CIN2), using a non-inferiority design. The primary objective is to demonstrate that ALA-PDT is non-inferior to LEEP with respect to key efficacy endpoints. Furthermore, the safety profiles, cervical tissue regeneration outcomes, and long-term prognoses of both treatment modalities will be comprehensively assessed. The results are anticipated to provide robust clinical evidence supporting ALA-PDT as a safer, less invasive, and function-preserving alternative for the management of HSIL/CIN2.

ELIGIBILITY:
Inclusion Criteria:

1. Female, 25-60 years, understands study procedures and consents to participate;
2. Colposcopy-guided cervical biopsy within 3 months showing HSIL/CIN2;
3. Provides written informed consent.

Exclusion Criteria:

1. Cytology showing ASC-H, HSIL, AGC, or AIS; or evidence of malignant cells on cytology/histology, or suspicion of malignancy or invasive cancer;
2. Colposcopy findings suggestive of invasive cancer or lesion extension to the vaginal wall;
3. Severe pelvic, cervical, or other gynecological inflammatory conditions identified clinically;
4. Undiagnosed vaginal bleeding;
5. Active allergic disease, porphyria, or history of allergy to the study drug or structurally similar agents;
6. Severe cardiovascular, neurological, psychiatric, endocrine, hepatic, or hematologic disorders; known immunodeficiency; long-term glucocorticoid or immunosuppressant use; active autoimmune disease; or other malignancies;
7. Pregnant or breastfeeding women;
8. History of hysterectomy, cervical cancer treatment, or cervical excision/ablation within 6 months (e.g., conization, LEEP, laser);
9. Use of interferon or antiviral therapy within 3 months;
10. Any other condition deemed unsuitable for participation by the investigator.

Ages: 25 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 560 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Lesion effective rate | 6 months
  Proportion of patients with LSIL or normal histopathology on colposcopy-guided cervical biopsy, assessed at 6 months post-treatment as the primary endpoint.

SECONDARY OUTCOMES:
Lesion effective rate | 2 years
  Proportion of patients with LSIL or normal histopathology on colposcopy-guided cervical biopsy, assessed at 12 and 24 months post-treatment.
HPV clearance rate | 2 years
  HPV clearance rates at 3, 6, 9, 12, and 24 months post-treatment
Lesion cure rate | 2 years
  Proportion of patients with normal colposcopy-guided cervical biopsy results and negative HPV

OTHER OUTCOMES:
Impact on cervical anatomy and function | 2 years
  Cervical length and function before and after treatment, and subsequent pregnancy outcomes in patients desiring fertility.
Adverse events | 2 years
  Record post-treatment adverse events including bleeding, infection, and pain.

CONTACTS AND LOCATIONS:
Locations (5):
- China (5):
  - Women's Hospital School Of Medicine Zhejiang University, Hangzhou, Zhejiang
  - First People's Hospital of Hangzhou, Hangzhou, Zhejiang
  - Hangzhou Linping District first People's Hospital, Hangzhou, Zhejiang
  - First Affiliated Hospital of Ningbo University, Ningbo, Zhejiang
  - Shaoxing People's Hospital, Shaoxing, Zhejiang

IPD SHARING:
Plan to Share IPD: No